CLINICAL TRIAL: NCT01008579
Title: Routine Use of Patient Reported Outcomes Among Older Adults at High Risk of Falls: A 12-Month Cohort Study
Brief Title: Assessing Patient Care Through Routine Use of Patient-Reported Outcomes
Status: Withdrawn | Type: Observational
Why Stopped: Redundant with another study
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Teresa Liu-Ambrose, Principal Investigator, University of British Columbia
Other Study IDs: H09-01655
Record Dates: First submitted 2009-11-04; First posted 2009-11-06 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Falls
Keywords: Patient Reported Outcome Measures; falls; older adults

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Patient reported outcome measures (PROMs) are assessments of health status or health-related quality of life. The EuroQol-5D (EQ5D) is an example of a generic instrument to assess health-related quality of life. The investigators will use the EQ5D in the Falls Prevention Clinic as part of routine clinical assessment at baseline, 6 months and 12 months to track patient care in a cohort of 300 older adults who are at high-risk of falls.

DETAILED DESCRIPTION:
1. Purpose: We will use the EQ5D in the Falls Prevention Clinic as part of routine clinical assessment at baseline, 6-months and 12-months to track patient care in a cohort of 300 older adults who are at high-risk of falls.
2. Objectives:

O1: Our primary objective is to use a routinely administered patient reported outcomes measure, the EuroQol-5D (EQ-5D), in older adults at high risk of falls to determine patients self-reported health status over a 12-month followup period.

O2: Our secondary objective is to develop an explanatory model and a predictive model of covariates that explain significant gains or losses in health related quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Referred to falls clinic for assessment by general practitioner or emergency department physician.
2. Index fall presentation not due to overwhelming force resulting in presentation to Emergency Department or general practitioner (including syncopal presentation, see below).
3. At least 70 years of age.
4. No progressive neurological disorder (e.g. Dementia, Parkinson's, Alzheimer's).
5. Community dwelling (within Vancouver and Burnaby only).
6. Mini Mental State Examination Score of at least 24.
7. Walk at least 3 meters.
8. Has at least one of the following 'high-risk' criteria:

   * At least one other non-syncopal fall in the past 12 months
   * PPA of at least 1.0 (using dominant score for strength test)
   * TUG of at least 15 seconds
9. Life expectancy of greater than 12 months as determined by the geriatrician.

Exclusion Criteria:

1. Any patients who do not meet the inclusion criteria specified above will be excluded from assessment at the Falls Prevention Clinic.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Falls Prevention Clinic
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-12; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karim Khan, Study Director — University of British Columbia; Teresa Liu-Ambrose, Study Director — University of British Columbia; Stirling Bryan, Principal Investigator — University of British Columbia
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada